CLINICAL TRIAL: NCT01478893
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Pharmacodynamics of Increasing Subcutaneous Doses of SEL-068 in Healthy Non-Smoker and Smoker Adults
Brief Title: Safety and Pharmacodynamics of SEL-068 Vaccine in Smokers and Non-Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Selecta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEL-068/101; 2011-003272-37 (EudraCT Number)
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Smoking Cessation
Keywords: nicotine vaccine; smoking vaccine; smoking cessation; SEL-068
MeSH Terms: conditions — Smoking Cessation | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SEL-068 (Experimental)
  Interventions: Biological: SEL-068
- Saline (Placebo Comparator)
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: SEL-068 — Sub-cutaneous injection, multiple dose
  Arms: SEL-068
Biological: Saline — Sub-cutaneous injection, multiple dose
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacodynamics of SEL-068. Increasing subcutaneous doses of SEL-068 will be administered to healthy non-smoker and smoker volunteers. The resulting safety profile and anti-nicotine antibody levels will be evaluated.

ELIGIBILITY:
Primary Inclusion Criteria:

* Healthy Smokers
* Healthy non-smokers
* Written informed consent

Primary Exclusion Criteria:

* Prior exposure to nicotine vaccines
* Female subjects of childbearing potential
* Current use of immunosuppressive agents
* History of or current autoimmune disorder of immunosuppressive condition (e.g. HIV infection)
* Concurrent participation or participation within 8 weeks prior to the initial study drug administration in a drug/device or biologic investigational research study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple subcutaneous injections of SEL-068 as assessed by frequency of vaccine related adverse events, graded by severity | 36 weeks

SECONDARY OUTCOMES:
Immunogenicity of SEL-068 by measuring anti-nicotine antibody titers by Enzyme-Linked Immunosorbent Assay (ELISA). | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva Vets, MD, Principal Investigator — SGS LSS Clinical Pharmacology Unit - Antwerpen
Locations (1):
- SGS LSS Clinical Pharmacology Unit, Antwerp, Belgium